CLINICAL TRIAL: NCT01927731
Title: Safety and Efficacy of Eltrombopag in Patients Undergoing Cord Blood or Haploidentical Bone Marrow Transplantation
Brief Title: Eltrombopag Olamine in Increasing Platelet Counts in Patients Undergoing Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0920; NCI-2013-02348 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0920 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Bone Marrow Transplantation Recipient; Cord Blood Transplant Recipient; Hematopoietic Cell Transplantation Recipient
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (cord blood transplant patients) (Experimental): Patients receive eltrombopag olamine PO QD for 60 days beginning on day -1.
  Interventions: Drug: Eltrombopag Olamine; Other: Laboratory Biomarker Analysis
- Arm II (haploidentical donor stem cell transplant patients) (Experimental): Patients receive eltrombopag olamine PO QD for 60 days beginning on day 5.
  Interventions: Drug: Eltrombopag Olamine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Eltrombopag Olamine — Given PO
  Other Names: Promacta; SB-497115-GR
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well eltrombopag olamine works in increasing platelet counts in patients undergoing transplant. Eltrombopag olamine may help platelet counts and the immune system recover from blood or bone marrow transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the rate of platelet engraftment by day 60 in patients undergoing cord blood transplant (CBT) or haploidentical donor stem cell transplantation treated with eltrombopag (eltrombopag olamine).

SECONDARY OBJECTIVES:

I. To assess safety of eltrombopag in this population. II. To assess neutrophil engraftment with eltrombopag in this population. III. To characterize immune reconstitution. IV. To assess overall survival (OS). V. To assess progression free survival (PFS). VI. To assess incidence of acute graft-versus-host disease (GVHD).

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (CORD BLOOD TRANSPLANT): Patients receive eltrombopag olamine orally (PO) once daily (QD) for 60 days beginning on day -1.

ARM II (HAPLOIDENTICAL DONOR STEM CELL TRANSPLANT): Patients receive eltrombopag olamine PO QD for 60 days beginning on day 5.

After completion of study treatment, patients are followed up at 1, 2, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a cord blood or haploidentical transplantation on any protocol or standard of care treatment plan.
* Age >/= 18.
* Females of child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization or breast-feeding must be willing to use an effective contraceptive measure until 30 days after the last dose of eltrombopag. Males who have had sexual contact with female of child-bearing potential must be willing to use contraceptive techniques until 30 days after the last dose of eltrombopag.
* Patient or patient's legal representative(s) is/are able to provide written informed consent to participate.

Exclusion Criteria:

* ALT and AST >/= 2.5 ULN.
* Serum direct bilirubin >/= 1 mg/dl (except Gilbert's syndrome or hemolysis).
* Patients of east Asian ancestry (Chinese, Japanese, or Korean Origin).
* Calculated creatinine clearance < 30ml./min. Creatinine clearance will be calculated using the MDRD method.
* Arterial or venous thrombosis in the last year except for line-related venous thrombosis more than 3 months ago.
* Positive beta HCG within 7 days prior to consent in female of child-bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uday Popat, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 2013 to November 2016. All participants were registered in University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Arm I (Cord Blood Transplant Patients) | Arm II (Haploidentical Donor Stem Cell Transplant Patients)
Started | 6 | 42
Completed | 3 | 32
Not Completed | 3 | 10
Not completed — Graft Failure | 1 | 2
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Cord Blood Transplant Patients) | Arm II (Haploidentical Donor Stem Cell Transplant Patients) | Total
Number analyzed (Participants) | 6 | 42 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 36 | 42
  >=65 years | 0 | 6 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 18 | 19
  Male | 5 | 24 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 8
  Not Hispanic or Latino | 5 | 35 | 40
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 42 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieved Platelet Engraftment Greater Than 50K/ul
Description: Number of participants that achieved platelet engraftment greater than 50K/ul 60 days post transplant.
Time Frame: Up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cord Blood Transplant Patients) | Arm II (Haploidentical Donor Stem Cell Transplant Patients)
Number analyzed (Participants) | 6 | 42
Participants | 3 | 30

2. Secondary Outcome: Overall Survival
Description: Number of participants that survived at one year post transplant.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cord Blood Transplant Patients) | Arm II (Haploidentical Donor Stem Cell Transplant Patients)
Number analyzed (Participants) | 3 | 32
Participants | 3 | 32

3. Secondary Outcome: Progression Free Survival
Description: Number of participants without disease progression at 1 year post transplant.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cord Blood Transplant Patients) | Arm II (Haploidentical Donor Stem Cell Transplant Patients)
Number analyzed (Participants) | 3 | 32
Participants | 3 | 30

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Arm I (Cord Blood Transplant Patients) | Arm II (Haploidentical Donor Stem Cell Transplant Patients)
All-Cause Mortality (participants affected / at risk) | 0/6 | 3/42
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/42
Other Adverse Events (participants affected / at risk) | 2/6 | 8/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cord Blood Transplant Patients) (N=6) | Arm II (Haploidentical Donor Stem Cell Transplant Patients) (N=42)
Sepsis (Infections and infestations) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Infections and infestations (Infections and infestations) | 2 | 2
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cord Blood Transplant Patients) (N=6) | Arm II (Haploidentical Donor Stem Cell Transplant Patients) (N=42)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2
Bronchial infection (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fever (General disorders) | 0 | 1
General disorders and administration site conditions (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Infections and infestations (Infections and infestations) | 0 | 8
Lethargy (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4
Nervous system disorders (Nervous system disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pleural infection (Infections and infestations) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Renal and urinary disorders (Renal and urinary disorders) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 4
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT01927731/Prot_SAP_000.pdf